CLINICAL TRIAL: NCT06086522
Title: A Phase I, Multicenter, Open-label, Dose Escalation and Dose Expansion Trial Evaluating the Safety, Pharmacodynamics, and Pharmacokinetics of Intravenous QN-302 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Trial to Evaluate Safety, PD & PK of IV Study Drug, QN-302, in Pts w/ Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qualigen Theraputics, Inc. (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 302P1V01
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation, Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Other): Starting dose in Phase 1a dose escalation
  Interventions: Drug: QN-302
- Cohort 2 (Other): 2nd cohort in Phase 1a dose escalation
  Interventions: Drug: QN-302

INTERVENTIONS:
Drug: QN-302 — Phase 1 dose-finding study, the study design is for QN-302 to be given once a week, intravenously over 60 min, on Day 1, Day 8, and Day 15 of a 28-Day cycle.

SUMMARY:
Goal: learn about QN-302 in patients with solid tumors (metastatic, or advanced cancer).

Main questions:

* What does the study drug do to human body (Pharmacodynamics [='PD'])
* What does the body do to study drug (how processed in body (Pharmacokinetics [='PK']) - Safety

Study drug by intravenous infusion ('IV') once weekly for 3 weeks every 4-week 'cycle.' Study treatment continues as long as patient and their study doctor agree that study treatment is in the best interest of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed locally advanced or metastatic solid carcinomas, who have had tumor progression after receiving all standard of care therapies or for which there is no approved therapy 2. Evaluable or measurable disease by RECIST 1.1

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine MTD | 18 months
  maximum tolerated dose identified from dose escalation cohorts
Establish RP2D | 24 months
  recommended Phase 2 dose identified from dose escalation cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Arshad, MD, Study Director — Qualigen Theraputics, Inc.
Locations (4):
- United States (4):
  - HonorHealth, Scottsdale, Arizona
  - Yale, New Haven, Connecticut
  - START Midwest, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided